CLINICAL TRIAL: NCT02689414
Title: A Study of Remote Ischaemic Preconditioning in Patients With Atherosclerosis Undergoing Vascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Jaak Kals, Clinic of Surgery, Department of Vascular Surgery, cardiovascular surgeon; MD-PhD, Tartu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16004
Record Dates: First submitted 2016-02-03; First posted 2016-02-24 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Abdominal Aortic Aneurysm; Peripheral Artery Disease; Carotid Artery Stenosis
Keywords: Atherosclerosis
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Peripheral Arterial Disease; Carotid Stenosis; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patient, patient's physician, surgeon, anaesthesiologist and everyone else in the surgical team were blinded to study intervention. Blinding was attained with manometer's scale covered. Second arterial stiffness measurement was carried out by a study member who did not know the patient's group affiliation.

ARMS (2):
- Remote ischaemic preconditioning (Experimental): Four episodes of 5 minutes of ischaemia are performed. Between all the episodes there is a 5-minute period of reperfusion.
  Interventions: Procedure: Remote ischaemic preconditioning
- Control to RIPC (Sham Comparator): Four episodes of 5 minutes during which the pressure in the cuff is equal to venous pressure are performed. Between all the episodes there is a 5-minute pause.
  Interventions: Procedure: Control to RIPC

INTERVENTIONS:
Procedure: Remote ischaemic preconditioning — Ischaemia is achieved by using a blood pressure cuff on an arm by raising the cuff pressure to 200 mm Hg or to a value that is 20 mm Hg greater than the patient's systolic blood pressure - if the patient's systolic blood pressure is more than 180 mm Hg. The intervention starts simultaneously with the induction of anaesthesia or a few minutes earlier.
  Other Names: RIPC
  Arms: Remote ischaemic preconditioning
Procedure: Control to RIPC — Venous pressure is achieved by using a blood pressure cuff on an arm by raising the cuff pressure to 10-20 mm Hg. The intervention starts simultaneously with the induction of anaesthesia or a few minutes earlier.
  Arms: Control to RIPC

SUMMARY:
The purpose of this study is to evaluate the effect of preoperative remote ischaemic preconditioning (RIPC) on organ damage and the functional characteristics of arteries in patients undergoing vascular surgery. In addition, we investigate the connection between RIPC and changes in the functional characteristics of arteries and low molecular weight metabolites.

ELIGIBILITY:
Inclusion Criteria:

* patients who are willing to give full informed consent for participation and
* who are undergoing open abdominal aortic aneurysm repair or
* who are undergoing endovascular aortic aneurysm repair or
* who are undergoing lower limb revascularization surgery or
* who are undergoing carotid endarterectomy

Exclusion Criteria:

* patients under age of 18
* patients who are pregnant
* patients with known malignancy during last 5 years
* patients with permanent atrial fibrillation or flutter
* patients with symptomatic upper limb atherosclerosis
* patients who require home oxygen therapy
* patients with eGFR < 30 ml/min/1.73 m2, measured preoperatively
* patients who have had myocardial infarction during last month
* patients who have had upper limb vein thrombosis
* patients who have undergone vascular surgery in the axillary region
* patients who are not able to follow the study regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-01; Primary Completion 2018-02-08 (Actual); Study Completion 2019-02

PRIMARY OUTCOMES:
Carotide-femoral pulse velocity | 24 h
  Measured with Sphygmocor XCEL
  * baseline characteristics are measured before surgery
  * measuring is repeated 24 h after surgery
Augmentation index | 24 h
  Measured with Sphygmocor XCEL
  * baseline characteristics are measured before surgery
  * measuring is repeated 24 h after surgery

SECONDARY OUTCOMES:
Cardiac markers | 24 h
  Troponin T, Creatine kinase-MB, N-terminal pro-brain natriuretic peptiide (NT-ProBNP).
Traditional biomarkers of renal function | 24 h
  Creatinine, Urea
Markers of inflammation and oxidative stress | 24 h
  Oxidized low-density lipoprotein (oxLDL), Interleukin-18 (IL-18), Myeloperoxidase (MPO), Isoprostane.
Duration of hospital stay | 30 days
Duration of intesive care unit stay | 30 days
Cardiac event | 10 days
  Myocardial infarction or cardiac arrest
Postoperative complications | 10 days
  Surgical wound infection or haematoma, Acute limb ischaemia, Acute deep vein thrombosis, Limb amputation, Pneumonia, Urinary tract infection.
1- year mortality | 1 year
Complications of remote ishcaemic preconditioning | 10 days
  Upper-extremity deep vein thrombosis, Acute upper limb ischaemia.
Novel biomarkers of renal function | 24 h
  Neutrophil gelatinase-associated lipocalin (NGAL), Liver-type fatty acid binding proteiin (L-FABP), Kidney Injury Molecule-1 (KIM-1), Cystatine C, β2 microglobulin (B2M),
Estimated glomerular filtration rate | 24 h
  eGFR
Low molecular-weight metabolites | 24 h
  * Acylcarnitines
  * Amino acids: leucine, ornithine, methionine, alanine, phenylalanine, valine, glutamate, tyrosine, glycine, arginine, citrulline, asparagine, aspartate, glutamine, histidine, lysine, proline, tryptophan, serine, threonine, cysteine and hydroxyproline.
  * Hydroxy acids: citrate, α-oxoglutarate, pyruvate, succinate, mallonic acid, β-hydroxybutyrate, cis-aconitic acid and oxaloacetate.
Arterial elasticity indices | 24 h
  Measured with HDI pulsewave CR-200
  * baseline characteristics are measured before surgery
  * measuring is repeated 24 h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Urmas Lepner, MD-PhD, Study Chair — Tartu University Hospital; Joel Starkopf, MD-PhD, Study Chair — Tartu University Hospital; Mihkel Zilmer, MD-PhD, Study Chair — University of Tartu; Jaak Kals, MD-PhD, Principal Investigator — Tartu University Hospital; Karl Kuusik, MD, Study Chair — University of Tartu; Teele Kepler, MD, Study Director — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Tartu County, Estonia

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250
- [Derived] Kasepalu T, Kuusik K, Lepner U, Starkopf J, Zilmer M, Eha J, Vahi M, Kals J. Remote ischaemic preconditioning influences the levels of acylcarnitines in vascular surgery: a randomised clinical trial. Nutr Metab (Lond). 2020 Sep 18;17:76. doi: 10.1186/s12986-020-00495-3. eCollection 2020. PMID 32968425
- [Derived] Kasepalu T, Kuusik K, Lepner U, Starkopf J, Zilmer M, Eha J, Vahi M, Kals J. Remote Ischaemic Preconditioning Reduces Kidney Injury Biomarkers in Patients Undergoing Open Surgical Lower Limb Revascularisation: A Randomised Trial. Oxid Med Cell Longev. 2020 Jan 23;2020:7098505. doi: 10.1155/2020/7098505. eCollection 2020. PMID 32047578
- [Derived] Kepler T, Kuusik K, Lepner U, Starkopf J, Zilmer M, Eha J, Lieberg J, Vahi M, Kals J. The Effect of Remote Ischaemic Preconditioning on Arterial Stiffness in Patients Undergoing Vascular Surgery: A Randomised Clinical Trial. Eur J Vasc Endovasc Surg. 2019 Jun;57(6):868-875. doi: 10.1016/j.ejvs.2018.12.002. Epub 2019 May 22. PMID 31126835